CLINICAL TRIAL: NCT02489968
Title: A Phase III, Randomised, Double-blind, Parallel Group, 24-week Study to Evaluate Efficacy and Safety of Once Daily Empagliflozin 10 mg and Linagliptin 5 mg Fixed Dose Combination Compared With Empagliflozin 10 mg Plus Placebo and a 52-week Study to Evaluate Efficacy and Safety of Once Daily Empagliflozin 25 mg and Linagliptin 5 mg Fixed Dose Combination Compared With Empagliflozin 25 mg Plus Placebo in Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control After 16-week Treatment With Empagliflozin (10 mg or 25 mg) Alone Once Daily.
Brief Title: Linagliptin as Add on Therapy to Empagliflozin 10 mg or 25 mg With Japanese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1275.13
Record Dates: First submitted 2015-05-27; First posted 2015-07-03 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- empagliflozin 10 mg + linagliptin 5 mg (Experimental): patient to receive a tablet containing low dose empagliflozin and linagliptin once daily
  Interventions: Drug: empagliflozin 10 mg + linagliptin 5 mg
- empagliflozin 10 mg (Experimental): patient to receive a tablet containing low dose empagliflozin once daily
  Interventions: Drug: empagliflozin 10 mg; Drug: Placebo
- empagliflozin 25 mg + linagliptin 5 mg (Experimental): patient to receive a tablet containing high dose empagliflozin and linagliptin once daily
  Interventions: Drug: empagliflozin 25 mg + linagliptin 5 mg
- empagliflozin 25 mg (Experimental): patients to receive a tablet containing high dose empagliflozin once daily
  Interventions: Drug: empagliflozin 25 mg; Drug: Placebo

INTERVENTIONS:
Drug: empagliflozin 10 mg + linagliptin 5 mg — empagliflozin low dose + linagliptin once daily
  Arms: empagliflozin 10 mg + linagliptin 5 mg
Drug: empagliflozin 10 mg — empagliflozin low dose once daily
  Arms: empagliflozin 10 mg
Drug: empagliflozin 25 mg + linagliptin 5 mg — empagliflozin high dose + linagliptin once daily
  Arms: empagliflozin 25 mg + linagliptin 5 mg
Drug: empagliflozin 25 mg — empagliflozin high dose once daily
  Arms: empagliflozin 25 mg
Drug: Placebo
  Arms: empagliflozin 10 mg; empagliflozin 25 mg

SUMMARY:
Two independent study parts (i.e. Part A and Part B) are included in this trial. Part A will evaluate empagliflozin 10 mg + linagliptin and Part B will evaluate empagliflozin 25 mg + linagliptin. All analyses will be carried out separately for these study parts. The objective of Part A is to investigate the efficacy, safety and tolerability of the fixed dose combination (FDC) of empagliflozin 10 mg / linagliptin 5 mg compared with empagliflozin 10 mg plus FDC matching placebo administered orally once daily for 24 weeks in Japanese patients with T2DM (Type 2 Diabetes Mellitus) who have insufficient glycaemic control after 16 weeks of treatment with empagliflozin 10 mg alone once daily. The study is designed to show superiority of the FDC of empagliflozin 10 mg / linagliptin 5 mg over empagliflozin 10 mg plus FDC matching placebo after 24 weeks of treatment. The objective of Part B is to investigate the efficacy, safety and tolerability of the FDC of empagliflozin 25 mg / linagliptin 5 mg compared with empagliflozin 25 mg plus FDC matching placebo administered orally once daily for 24 weeks in Japanese patients with T2DM who have insufficient glycaemic control after 16 weeks of treatment with empagliflozin 25 mg alone once daily. The study is designed to show superiority of the FDC of empagliflozin 25 mg / linagliptin 5 mg over empagliflozin 25 mg plus FDC matching placebo after 24 weeks of treatment. The 24 week treatment period will be followed by a 28 week extension treatment period to evaluate further efficacy and safety up to 52 weeks.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of type 2 diabetes prior to informed consent
* Male and female patients on diet and exercise regimen for at least 12 weeks prior to informed consent who are:

  * drug-naïve, defined as no antidiabetic drugs for at least 12 weeks prior to informed consent or,
  * pre-treated with one oral antidiabetic drug (for sulfonylurea, with up to half of the maximum approved dose) on stable dosage for at least 12 weeks prior to the informed consent (for thiazolidinedione, therapy has to be unchanged for at least 18 weeks prior to the informed consent). Individual antidiabetic drug will have to be discontinued at Visit 1.
* haemoglobin A1c (HbA1c) at Visit 1 (screening)

  * for patients without antidiabetic therapy : HbA1c >=8.0 to =<10.5%
  * for patients with one oral antidiabetic drug : HbA1c >=7.5 to =<10.5%
* HbA1c >=7.5 to =<10.0% at Visit 4 for randomisation into the double blind treatment period

Exclusion criteria:

* Uncontrolled hyperglycaemia with a glucose level >270 mg/dL (>15.0 mmol/L) during the open label stabilisation period and placebo run in period
* Impaired renal function, defined as estimated glomerular filtration rate (eGFR) <45 mL/min/1.73m2 (modification of diet in renal disease (MDRD) formula)
* Acute coronary syndrome, stroke or transient ischemic attack (TIA) within 12 weeks prior to informed consent
* Indication of liver disease, defined by serum levels of either alanine transaminase (ALT), aspartate transaminase (AST), or alkaline phosphatase (ALP) above 3 x upper limit of normal (ULN)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2017-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (83):
- Japan (83):
  - Tokai Memorial Hospital, Aichi, Kasugai
  - Japan Organization of Occupational Health and Safety Chubu Rosai Hospital, Aichi, Nagoya
  - Tokuyama Clinic, Chiba, Chiba
  - Matsuyama Shimin Hospital, Ehime, Matsuyama
  - Tanaka Int. Clinic, Ehime, DIA Med.,CV Med., Ehime, Niihama
  - Murakami Memorial Hp., Ehime, I.M., Ehime, Saijo
  - Kunisaki Makoto Clinic, Fukuoka, I.M./CV Med., Fukuoka, Fukuoka
  - Fukuoka Shin Mizumaki Hospital, Fukuoka, Onga
  - Shin Yukuhashi Hospital, Fukuoka, Yukuhashi
  - Hashimoto I.M., Gifu, I.M., Gifu, Gifu
  - Kikuchi Naika Clinic, Gunma, I.M., Gunma, Maebashi
  - Hasegawa Internal Medicine Clinic, Hokkaido, Chitose
  - Ebetsu Internal Medicine Clinic, Hokkaido, Ebetsu
  - Hakodate Koseiin Hakodate Central General Hospital, Hokkaido, Hakodate
  - Iida Medical Clinic, Hokkaido, Hakodate
  - Kurihara Clinic, Hokkaido, Sapporo
  - Uehara Clinic, Hokkaido, Sapporo
  - Manda Memorial Hospital, Hokkaido, Sapporo
  - Sapporo Diabetes, Thyroid Clinic, Hokkaido, Sapporo
  - Japan Community Health Care Organization Hokkaido Hospital, Hokkaido, Sapporo
  - Ashiya Municipal Hospital, Hyogo, Ashiya
  - Itabashi DIA Med. and DERM Clinic, Ibaraki, I.M., Ibaraki, Koga
  - Namegata District General Hospital, Ibaraki, Namegata
  - Hokuriku Hp., Ishikawa, I.M., Ishikawa, Kanazawa
  - Oikawa Clinic, Iwate, Morioka
  - Hirano Medical Clinic, Iwate, Morioka
  - Iwamoto Clinic, Kagawa, DIAB I.M., Kagawa, Zentsuji
  - Tenpozan Clinic of I.M., Kagoshima, I.M., Kagoshima, Kagoshima
  - Hayashi DIA Clinic, Kanagawa, DIA Tract Med.·I.M., Kanagawa, Chigasaki
  - Takai Naika Clinic, Kanagawa, Kamakura
  - Nagatsuta Family Clinic, Kanagawa, I.M., Kanagawa, Yokohama
  - Motomachi Takatsuka Naika Clinic, Kanagawa, I.M., Kanagawa, Yokohama
  - Yokohama Minoru Clinic, Kanagawa, Yokohama
  - Morinagaueno clinic, Kumamoto, Digestive Tract I.M., Kumamoto, Kumamoto
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Jinnouchi Clinic Diabetes Care Center, Kumamoto, Kumamoto
  - Kajiyama Clinic, Kyoto, I.M., Kyoto, Kyoto
  - Matsumoto Nakagawa Hospital, Nagano, Matsumoto
  - Ota DIA I.M. Clinic, Nagano, I.M., Nagano, Nagano
  - Saiseikai Niigata Daini Hp., Niigata, METAB ENDO, Niigata, Niigata
  - Tsuyama Chuo Hospital, Okayama, Tsuyama
  - Yaesu Clinic, Okinawa, I.M., Okinawa, Naha
  - Tanaka Clinic, Okinawa, I.M., Okinawa, Tomigusuku
  - AMC Nishi-umeda Clinic, Osaka
  - Shiraiwa Medical Clinic, Osaka, I.M., Osaka
  - Umeda Oak Clinic, Osaka, I.M., Osaka, Osaka
  - Kinugawa CARDIOL Clinic, Osaka, I.M., Osaka, Osaka
  - Ikeoka Clinic, Osaka, I.M., Osaka, Osaka
  - Nanko Clinic, Osaka, I.M., Osaka, Osaka
  - OCROM Clinic, Osaka, Suita
  - Saga Memorial Hospital, Saga, Saga
  - Odayaka Life Naika Clinic, Saitama, I.M., Saitama, Koshigaya
  - Medical corporation Chisei-kai Watanabe clinic, Saitama, Okegawa
  - Medical Corporation Toujinkai Sakado Central Hospital, Saitama, Sakado
  - SAINO Clinic,, Saitama, Tokorozawa
  - Hamamatsu Rosai Hospital, Shizuoka, Hamamatsu
  - Plumeria Clinic, Shizuoka, I.M., Shizuoka, Shizuoka
  - Wakakusa Clinic, Tochigi, I.M., Tochigi, Shimotsuke
  - Kanda Clinic, Tokyo, I.M., Tokyo
  - Nihonbashi Sakura Clinic, Tokyo, Chuo-ku
  - Fukuwa Clinic, Tokyo, Chuo-ku
  - Nihonbashi Enomoto Internal Medicine, Tokyo, Chuo-ku
  - Tokyo-Eki Center-building Clinic, Tokyo, Chuo-ku
  - Tokyo Center Clinic, Tokyo, Chuo-ku
  - Hosono Clinic, Tokyo, Chuo-ku
  - AGE Makita Medical Clinic, Tokyo, Chuo-ku
  - Kasai Diabetes Clinic, Tokyo, Edogawa-ku
  - New Medical Research System Clinic, Tokyo, Hachioji
  - Medical Corporation Keikokai P1-Clinic, Tokyo, Hachioji
  - Minamino Heart Clinic, Tokyo, Hachioji
  - Shinkoiwa Ekimae Sougou Clinic, Tokyo, Katushika-ku
  - Musashino Polyclinic, Tokyo, Kiyose
  - Pedi Shiodome Clinic, Tokyo, Minato-ku
  - Shinagawa East one Medical Clinic, Tokyo, Minato-ku
  - Shimamura Kinen Hospital, Tokyo, Nerima-ku
  - Kenkoukan Suzuki Clinic, Tokyo, Ota-ku
  - Honda Hidehiko Clinic, Tokyo, Ota-ku
  - Sakayori Clinic, Tokyo, Shinagawa-ku
  - Miho Clinic, Tokyo, Shinagawa-ku
  - ToCROM Clinic, Tokyo, Shinjuku-ku
  - Ikebukuro Metropolitan Clinic, Tokyo, Toshima-ku
  - Fujikoshi Hp., Toyama, I.M., Toyama, Toyama
  - Clinic Sugiyama, Yamagata, I.M., Yamagata, Yamagata

REFERENCES:
- [Derived] Kaku K, Haneda M, Tanaka Y, Lee G, Shiki K, Miyamoto Y, Solimando F, Lee J, Lee C, George J. Linagliptin as add-on to empagliflozin in a fixed-dose combination in Japanese patients with type 2 diabetes: Glycaemic efficacy and safety profile in a two-part, randomized, placebo-controlled trial. Diabetes Obes Metab. 2019 Jan;21(1):136-145. doi: 10.1111/dom.13496. Epub 2018 Sep 6. PMID 30091172

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 880 subjects started the open label period
Groups:
- Empagliflozin 10 mg OL: Patients were administered empagliflozin 10 milligram (mg) tablets, orally with water, once daily for 16-weeks of open-label stabilisation period.
- Empagliflozin 25 mg OL: Patients were administered empagliflozin 25 mg tablets, orally with water, once daily for 16-weeks of open-label stabilisation period.
- Empagliflozin 10 mg + Linagliptin 5 mg: Patients who received empagliflozin 10 mg during open-label stabilisation period were randomized to receive a fixed dose combination (FDC) tablet of empagliflozin 10 mg and linagliptin 5 mg along with a matching placebo of empagliflozin 10 mg, orally with water, once daily for 24-weeks of double-blind treatment period.
- Empagliflozin 10 mg + Placebo: Patients who received empagliflozin 10 mg during open-label stabilisation period were randomized to receive empagliflozin 10 mg along with a matching placebo of the FDC tablet of empagliflozin 10 mg and linagliptin 5 mg, orally with water, once daily for 24-weeks of double-blind treatment period.
- Empagliflozin 25 mg + Linagliptin 5 mg: Patients who received empagliflozin 25 mg during open-label stabilisation period were randomized to receive a FDC tablet of empagliflozin 25 mg and linagliptin 5 mg along with a matching placebo of empagliflozin 25 mg, orally with water, once daily for 52-weeks of double-blind treatment period.
- Empagliflozin 25 mg + Placebo: Patients who received empagliflozin 25 mg during open-label stabilisation period were randomized to receive empagliflozin 25 mg along with a matching placebo of the FDC tablet of empagliflozin 25 mg and linagliptin 5 mg, orally with water, once daily for 52-weeks of double-blind treatment period.
Period: Open-label Treatment Period
Arm/Group | Empagliflozin 10 mg OL | Empagliflozin 25 mg OL | Empagliflozin 10 mg + Linagliptin 5 mg | Empagliflozin 10 mg + Placebo | Empagliflozin 25 mg + Linagliptin 5 mg | Empagliflozin 25 mg + Placebo
Started | 439 | 440 (1 subject did not receive treatment and hence excluded. Started represents treated numbers.) | 0 | 0 | 0 | 0
Completed | 215 | 232 | 0 | 0 | 0 | 0
Not Completed | 224 | 208 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 14 | 7 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 7 | 0 | 0 | 0 | 0
Not completed — Other than specified above | 204 | 189 | 0 | 0 | 0 | 0
Period: Double-blind Treatment Period
Arm/Group | Empagliflozin 10 mg OL | Empagliflozin 25 mg OL | Empagliflozin 10 mg + Linagliptin 5 mg | Empagliflozin 10 mg + Placebo | Empagliflozin 25 mg + Linagliptin 5 mg | Empagliflozin 25 mg + Placebo
Started | 0 | 0 | 107 | 108 | 116 | 116
Completed | 0 | 0 | 105 | 100 | 110 | 108
Not Completed | 0 | 0 | 2 | 8 | 6 | 8
Not completed — Adverse Event | 0 | 0 | 2 | 6 | 4 | 5
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 2
Not completed — Other than specified above | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Open-label full analysis set (OLFAS) consisted of all patients in the open-label period who received at least 1 dose of open-label study drug during the trial and had a pre-treatment Glycated haemoglobin A1c (HbA1c) assessment and at least 1 on-treatment HbA1c assessment during the open-label part of the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin 10 mg OL | Empagliflozin 25 mg OL | Total
Number analyzed (Participants) | 435 | 433 | 868
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (10.2) | 57.5 (10.0) | 57.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 124 | 235
  Male | 324 | 309 | 633

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycated Haemoglobin A1c (HbA1c) (%) From Baseline After 24 Weeks of Treatment
Description: Change from baseline in HbA1c (%) after 24 weeks of treatment with double-blind trial medication. Change was calculated as: HbA1c value at 24-week - HbA1c value at baseline, for each patient. Baseline was defined as the last observation before the first intake of double-blind randomised trial medication. Statistical analysis presented is based on a restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) approach. Full Analysis Set (Observed Cases) [FAS (OC)]: This analysis set consisted of all patients who were randomised and treated with at least 1 dose of trial drug during the double-blind part of the trial and who had a baseline HbA1c assessment and at least 1 on-treatment HbA1c assessment during the 24-week double-blind part of the trial. Observed cases analysis included only the available data that were observed while patients were on treatment, i.e., excluding the missing data.
Time Frame: Baseline and 24 week
Population: FAS (OC)
Measure: Least Squares Mean (Standard Error); unit: Percentage (%)
Arm/Group | Empagliflozin 10 mg + Linagliptin 5 mg | Empagliflozin 10 mg + Placebo | Empagliflozin 25 mg + Linagliptin 5 mg | Empagliflozin 25 mg + Placebo
Number analyzed (Participants) | 103 | 96 | 111 | 108
Percentage (%) | -0.94 (0.05) | -0.12 (0.06) | -0.91 (0.05) | -0.33 (0.05)
Statistical Analysis 1: Comparison: Empagliflozin 10 mg + Linagliptin 5 mg vs Empagliflozin 10 mg + Placebo; Test type: Superiority or Other; p < 0.0001, REML based MMRM; Model including baseline HbA1c, treatment, baseline renal function, prior use of antidiabetic drug, visit, and visit by treatment interaction; Adjusted mean difference = -0.82, 95% CI 2-sided [-0.97 to -0.67], Standard Error of Mean 0.08 — Adjusted mean difference: Change in HbA1c in (empagliflozin 10 mg + linagliptin 5 mg) - change in HbA1c in (empagliflozin 10 mg + placebo)
Statistical Analysis 2: Comparison: Empagliflozin 25 mg + Linagliptin 5 mg vs Empagliflozin 25 mg + Placebo; Test type: Superiority or Other; p < 0.0001, REML based MMRM; [statistical method as in outcome 1, analysis 1]; Adjusted mean difference = -0.59, 95% CI 2-sided [-0.73 to -0.45], Standard Error of Mean 0.07 — Adjusted mean difference: Change in HbA1c in (empagliflozin 25 mg + linagliptin 5 mg) - change in HbA1c in (empagliflozin 25 mg + placebo)

ADVERSE EVENTS:
Time Frame: From first drug administration till two weeks after last drug administration; up to 72 weeks (including 16 weeks open-label, 2 weeks run-in period and 52 weeks double-blind treatment period).
Description: All patients who were randomised and treated with at least 1 dose of trial drug during open-label and double-blind part of the trial. Adverse events were coded using the MedDRA coding system version 19.1 (Week 24 analysis) and version 20.0 (Week 52 analysis).
Arm/Group | Empagliflozin 25 mg + Linagliptin 5 mg | Empagliflozin 10 mg + Linagliptin 5 mg | Empagliflozin 25 mg + Placebo | Empagliflozin 10 mg + Placebo | Empagliflozin 25 mg OL | Empagliflozin 10 mg OL
Serious Adverse Events (participants affected / at risk) | 6/116 | 1/107 | 8/116 | 4/108 | 11/440 | 9/439
Other Adverse Events (participants affected / at risk) | 54/116 | 24/107 | 51/116 | 36/108 | 131/440 | 120/439
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 25 mg + Linagliptin 5 mg (N=116) | Empagliflozin 10 mg + Linagliptin 5 mg (N=107) | Empagliflozin 25 mg + Placebo (N=116) | Empagliflozin 10 mg + Placebo (N=108) | Empagliflozin 25 mg OL (N=440) | Empagliflozin 10 mg OL (N=439)
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Diabetic gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lateral medullary syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Torus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis E (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 25 mg + Linagliptin 5 mg (N=116) | Empagliflozin 10 mg + Linagliptin 5 mg (N=107) | Empagliflozin 25 mg + Placebo (N=116) | Empagliflozin 10 mg + Placebo (N=108) | Empagliflozin 25 mg OL (N=440) | Empagliflozin 10 mg OL (N=439)
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 35 | 30
Blood ketone body increased (Investigations) | 16 | 2 | 9 | 11 | 40 | 26
Weight decreased (Investigations) | 2 | 0 | 7 | 1 | 10 | 16
Viral upper respiratory tract infection (Infections and infestations) | 31 | 16 | 34 | 24 | 46 | 47
Periodontitis (Infections and infestations) | 3 | 0 | 6 | 1 | 2 | 2
Constipation (Gastrointestinal disorders) | 5 | 2 | 6 | 0 | 11 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 3 | 2 | 3 | 5 | 2
Contusion (Injury, poisoning and procedural complications) | 4 | 3 | 6 | 1 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.